1007779

**Sponsor Name:** Theracos Sub, LLC

Protocol Number and Title: A Phase 3, Randomized, Double-Blind, Active-

Controlled Study to Evaluate the Effects of Bexagliflozin versus Sitagliptin in Subjects with Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control by Metformin

Protocol Version and Date: Version 2.0, 06 April 2017

INC Research Project Code: 1007779

Author(s): Lu Wang, Biostatistician II

SAP Version: Version 1.0

SAP Version Date: 28-Feb-2018

#### Notice of Confidential and Proprietary Information:

The information contained in this document is confidential belonging to Theracos Sub, LLC. Acceptance of this document constitutes agreement by the recipient that no information contained herein will be published or disclosed without prior written authorization from an official of Theracos Sub, LLC. However, this document may be disclosed to appropriate Institutional Review Board and Ethics Committees or duly authorized representatives of a national regulatory authority under the condition that they are requested to keep it confidential. In the event of an actual or suspected breach of this obligation, INC Research should be notified promptly.

Version 1.0

THR-1442-C-423

1007779

# **Revision History**

| Version # Date (dd-mmm-yyyy) | | Document Owner | Revision Summary |
|---|---|---|---|
| Version 0.1 | 24-Jan-2018 | Lu Wang | Initial Release Version |
| Version 0.2 | 06-Feb-2018 | Lu Wang | Update to Address Sponsor<br>Comments |
| Version 1.0 | 28-Feb-2018 | Lu Wang | Update to Address Sponsor<br>Comments |

I confirm that I have reviewed this document and agree with the content.

| APPROVALS | |
|---------------------------------------|--------------------|
| INC Research | |
| Lu Was | 0t-1Na4-2018 |
| Lead Biostatistician | Date (dd-Mmm-yyyy) |
| Lu Wang | |
| Biostatistician II | |
| 40 | 05-Mar-2018 |
| Senior Reviewing Biostatistician | Date (dd-Mmm-yyyy) |
| Fang Zhu | |
| Senior Biostatistician, Biostatistics | |
| Theracos Sub, LLC | |
| Mundi Has | 02- Mar - 2018 |
| Sponsor Contact | Date (dd-Mmm-yyyy) |
| Yuan-Di Halvorsen | |
| Program Manager for Theracos Sub, LLC | |

# **TABLE OF CONTENTS**

| 1. G | LOSSARY OF ABBREVIATIONS | 8 |
|------------------------|------------------------------------|----|
| 2. Pl | URPOSE | 11 |
| 2.1. | Responsibilities | 11 |
| 2.2. | Timings of Analyses | 11 |
| 3. <b>S</b> 7 | TUDY OBJECTIVES | 12 |
| 3.1. | Primary Objective | 12 |
| 3.2. | Key Secondary Objectives | 12 |
| 3.3. | Safety Objectives | 12 |
| 3.4. | Brief Description | 13 |
| 3.5.<br>3.5.1<br>3.5.2 | | 14 |
| 3.6. | Determination of Sample Size | 14 |
| 3.7.<br>3.7.1<br>3.7.2 | | 15 |
| 3.8. | Administration of Study Medication | 15 |
| 3.9. | Study Procedures and Flowchart | 16 |
| 4. El | NDPOINTS | 19 |
| 4.1. | Primary Efficacy Endpoint | 19 |
| 4.2. | Secondary Efficacy Endpoints | 19 |
| 4.3. | Safety Endpoints | 19 |
| 5. AI | NALYSIS SETS | 20 |

| 5.1. | Screened Analysis Set | 20 |
|-----------------|-------------------------------------------------|-----|
| 5.2. | Safety Analysis Set | 20 |
| 5.3. | Intention to Treat Analysis Set | 20 |
| 5.4. | Per Protocol Analysis Set | 20 |
| 5.5. | Protocol Deviations | 20 |
| | | 0.0 |
| 6. | GENERAL ASPECTS FOR STATISTICAL ANALYSIS | 22 |
| 6.1. | General Methods | 22 |
| 6.2. | Key Definitions | 22 |
| 6.2 | | |
| 6.2 | | |
| 6.2 | .3. Study Day | 23 |
| 6.2 | | |
| 6.2 | | |
| 6.3. | Missing Data | 22 |
| 0.3. | wissing Data | 23 |
| 6.4. | Analysis Visit Windows | 23 |
| 6.5. | Pooling of Centers | 24 |
| | DEMOGRAPHIC, OTHER BASELINE CHARACTERISTICS AND | 0.5 |
| MED | ICATION | 25 |
| 7.1. | Subject Disposition and Withdrawals | 25 |
| 7.2. | Subject Eligiblity and Protocol Deviations | 25 |
| 7.3. | Demographic and Other Baseline Characteristics | 25 |
| 7.4. | Medical History | |
| / • <b>-1</b> • | modical riistory | 20 |
| 7.5. | Medication | 26 |
| 7.5 | .1. Prior Medication | 26 |
| 7.5 | .2. Concomitant Medication | 27 |
| <b>8.</b> | EFFICACY | 28 |
| 8.1. | Primary Efficacy Endpoint and Analysis | 28 |
| 8.1 | | |
| O. 1 | | |

| 8 | .1.2. | Sensitivity Analyses | 29 |
|---|---|---|---|
| 8 | .1.3. | Subgroups | 32 |
| 8.2. | Sec | condary Efficacy Endpoint(s) and Analyses | 32 |
| | .2.1. | Change in FPG in the bexagliflozin group vs. the sitagliptin group at week 24 | |
| _ | .2.2. | Change in body weight in subjects with baseline body mass index (BMI) ≥ 25 kg | ן/m² in |
| th | ne bexa | gliflozin group vs. the sitagliptin group at week 24 | 33 |
| | .2.3. | Change in SBP in the bexagliflozin group vs. the sitagliptin group at week 24 | |
| | .2.4. | Sensitivity analysis | 33 |
| | .3.1. | Change from baseline in HbA1c, SBP, Body weight, and in FPG over time | |
| 8 | .3.2. | Proportions of subjects with HbA1c of < 7% over time | 34 |
| 9. | SAFI | ETY | 35 |
| 9.1. | Ext | tent of Exposure | 35 |
| 9.2. | Tro | eatment Compliance | 26 |
| 9.2. | ire | aunent Compilance | 30 |
| 9.3. | Ad | verse Events | 36 |
| - | .3.1. | Derived Data | |
| | .3.2. | Data Summarization | |
| 9 | .3.3. | AE of Special Interest | 38 |
| 9.4. | Lal | ooratory Evaluations | 40 |
| 9.5. | Vita | al Signs | 43 |
| 9.6. | Ele | ctrocardiogram | 43 |
| 9.7. | Ph | ysical Examination | 43 |
| 10. | IN <sup>.</sup> | TERIM ANALYSES | 45 |
| 100 | | | |
| 11. | DA | ATA AND SAFETY MONITORING BOARD | 45 |
| 12. | C⊦ | HANGE FROM ANALYSIS PLANNED IN PROTOCOL | 45 |
| 14. | 0. | | |
| 13. | RE | FERENCE LIST | 46 |
| 14. | PR | ROGRAMMING CONSIDERATIONS | 47 |
| 14.1 | | neral Considerations | |
| 14.2 | . Tal | ole, Listing, and Figure Format | 48 |

# Version 1.0

# THR-1442-C-423

| 14.2.<br>14.2.<br>14.2.<br>14.2.<br>14.2.<br>14.2. | <ol> <li>Display Titles</li> <li>Column Headers</li> <li>Body of the Data Display</li> </ol> | 48<br>49<br>49<br>49 |
|---|---|---|
| 15. | QUALITY CONTROL | 52 |
| 16. | INDEX OF TABLES | 53 |
| 17. | INDEX OF FIGURES | 53 |
| 18. | INDEX OF LISTINGS | 53 |
| 19. | MOCK-UPS | 53 |
| 20. | APPENDICES | 53 |

# 1. GLOSSARY OF ABBREVIATIONS

| Abbreviation | Description |
|--------------|-------------------------------------------|
| AE | Adverse Event |
| ANCOVA | Analysis of Covariance |
| ATC | Anatomical Therapeutic Chemical |
| BMI | Body Mass index |
| ВР | Blood Pressure |
| CEC | Cardiovascular Endpoint Committee |
| CI | Confidence Interval |
| CRF | Case Report Form |
| DKA | Diabetic Ketoacidosis |
| dL | Deciliter |
| DSMB | Data and Safety Monitoring Board |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| eGFR | Estimating Glomerular Filtration Rate |
| FPG | Fasting Plasma Glucose |
| GEE | Generalized Estimating Equation |
| GMI | Genital Mycotic Infection |
| HbA1c | Hemoglobin A1c |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonization |
| ITT | Intention to Treat |
| IWRS | Interactive Web Randomization System |
| LDL-C | Low Density Lipoprotein Cholesterol |
| LOCF | Last Observation Carried Forward |
| LS | Least Squares |
| MACE | Major Adverse Cardiovascular Event |

Version 1.0

THR-1442-C-423

| Abbreviation | Description |
|---|---|
| MAR | Missing at Random |
| MCAR | Missing Completely at Random |
| MCMC | Monte Carlo Markov Chain |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | Milligram |
| mL | Milliliter |
| MMRM | Mixed Model Repeated Measures |
| MNAR | Missing not at Random |
| N/A | Not Applicable |
| Na | Sodium |
| PP | Per Protocol |
| PR | Time from the beginning of the P wave to the beginning of the QRS complex in electrocardiogram |
| PT | Preferred Term |
| Q1 | 1 <sup>st</sup> Quartile |
| Q3 | 3 <sup>rd</sup> Quartile |
| QRS | Graphical deflections corresponding to ventricular depolarization in a typical electrocardiogram |
| QTc | Time between the start of the Q wave and the end of the T wave in the ECG, corrected for heart rate |
| RR | Time between the start of one R wave and the start of the next R wave in the ECG |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SBP | Systolic Blood Pressure |
| SD | Standard Deviation |
| SE | Standard Error |
| SI | Standard International System of Units |
| SMBG | Self-Monitored Blood Glucose |
| SOC | System Organ Class |

Version 1.0

THR-1442-C-423

| Abbreviation | Description |
|--------------|-------------------------------------------|
| SOP | Standard Operating Procedure |
| T2DM | Type 2 Diabetes Mellitus |
| TEAE | Treatment-emergent Adverse Event |
| TLF | Table, Listing And Figure |
| UACR | Urine Albumin To Creatinine Ratio |
| UTI | Urinary Tract Infection |
| WBC | White Blood Cell |
| WHO-DD | World Health Organization Drug Dictionary |

1007779

#### 2. PURPOSE

The purpose of this statistical analysis plan (SAP) is to ensure that the data listings, summary tables and figures which will be produced, and the statistical methodologies that will be used, are complete and appropriate to allow valid conclusions regarding the study objectives.

# 2.1. RESPONSIBILITIES

Theracos has designed the study protocol and is responsible for the conduct of the study. INC Research is responsible for the development and validation of a clinical database using MediData RAVE platform.

INC Research will perform the statistical analyses and are responsible for the production and quality control of all tables, figures and listings (TLFs).

Adverse events that have met the seriousness criteria defined in the protocol are reported on the serious adverse event (SAE) forms using the MediData RAVE platform. An SAE case consists of the information reported in the SAE forms, subject characteristics documented in the case report forms, and additional source data such as hospital discharge summaries. Each SAE case is recorded in a validated ARGUS database which is managed by Covance. Any discrepancies in critical data fields of each SAE will be reconciled between the AUGUS and THR-1442-C-423 clinical database prior to database lock. The SAE coding, analyses and summaries are based on the final study data recorded in the clinical database. Detailed serious adverse event follow-up data will be reported from the ARGUS database and are not included in this report.

Theracos will perform review of all tables, figures and listings before the finalization.

#### 2.2. TIMINGS OF ANALYSES

The final analysis of safety and efficacy is planned after all subjects complete the planned 24 weeks of blinded study treatment and the subsequent follow-up period or terminate early from the study.

# 3. STUDY OBJECTIVES

# 3.1. PRIMARY OBJECTIVE

To demonstrate that bexagliflozin is non-inferior to sitagliptin by evaluating the treatment effect on hemoglobin A1c (HbA1c) reduction at week 24 in subjects whose type 2 diabetes mellitus (T2DM) is not adequately controlled by metformin.

## 3.2. KEY SECONDARY OBJECTIVES

The key secondary efficacy objectives of this study are:

- To evaluate the treatment effect of bexagliflozin vs. sitagliptin on the change in fasting plasma glucose (FPG) at week 24.
- To evaluate the treatment effect of bexagliflozin vs. sitagliptin on the change in body weight in subjects with baseline body mass index (BMI) ≥ 25 kg/m² at week 24.
- To evaluate the treatment effect of bexagliflozin vs. sitagliptin on the change in systolic blood pressure (SBP) in subjects at week 24.

The other exploratory secondary efficacy objectives are:

- To assess the treatment effect of bexagliflozin vs. sitagliptin on the change in the proportion of subjects achieving HbA1c < 7.0 % over time.
- To assess the treatment effect of bexagliflozin vs. sitagliptin on the change in HbA1c over time.
- To assess the treatment effect of bexagliflozin vs. sitagliptin on the change in FPG over time.
- To assess the treatment effect of bexagliflozin vs. sitagliptin on the change in body weight over time.
- To assess the treatment effect of bexagliflozin vs. sitagliptin on the change in SBP over time.

# 3.3. SAFETY OBJECTIVES

• To compare the effects of bexagliflozin with sitagliptin on the incidence of adverse events (AE) of interest. AE of interest are urinary tract infections (UTI) including urosepsis and pyelonephritis, genital mycotic infections (GMI), diuretic

1007779

effects including hypovolemia, hypotension episodes, hypoglycemia, hepatotoxicity, major adverse cardiovascular events (MACE), falls and fractures, malignancies, hypersensitivity reactions, acid-base disorders including diabetic ketoacidosis (DKA), amputations, pancreatitis, and renal failure events.

• To compare the effects of bexagliflozin with sitagliptin on general safety assessments including treatment emergent AEs, clinical laboratory findings, 12-lead electrocardiograms (ECG) parameters, physical examinations, vital signs including orthostatic blood pressure (BP), and use of concomitant medications.

#### 3.4. BRIEF DESCRIPTION

THR-1442-C-423 is a phase 3, multi-center, randomized, double-blind, parallel-group study and aims to demonstrate that bexagliflozin is non-inferior to sitagliptin as an add-on therapy in subjects whose T2DM is not adequately controlled by metformin treatment. A total of 374 subjects are planned to be randomized in a ratio of 1:1 to receive once daily treatment of bexagliflozin tablets, 20 mg, with sitagliptin tablets, placebo (Group 1) or bexagliflozin tablets, placebo, with sitagliptin tablets, 100 mg (Group 2) for 24 weeks in an outpatient setting. The main eligibility criteria include 1) male or female subjects with T2DM and 2) screening HbA1c between 7.0% and 11% (inclusive).

Qualified subjects must have taken metformin at a stable dose of  $\geq$  1500 mg/day in addition to diet and exercise counseling for at least 8 weeks prior to screening. Study subjects will continue taking open-labeled metformin during the entire study.

All eligible subjects will start a single-blind run-in period by taking placebo bexagliflozin and placebo sitagliptin once daily for one week. Subjects who meet all inclusion criteria and no exclusion criteria after completion of the run-in period will be eligible for randomization and receive investigational products.

During the treatment period, subjects will receive once daily sitagliptin tablets 100 mg with dummy placebo bexagliflorzin, or bexagliflozin tablets 20 mg with dummy placebo sitagliptin tablets, for 24 weeks. Each subject will be instructed to return to the clinic at weeks 6, 12, 18, and 24 for efficacy assessment and safety monitoring. Subjects will return to the clinic for a follow-up exit visit at week 26 or 2 weeks after last dose of study drug if subjects early terminate prior to week 24.

#### 3.5. SUBJECT SELECTION

The study population will include approximately 374 subjects whose T2DM is inadequately controlled by metformin and who meet all of the inclusion criteria and none of the exclusion criteria. Clinical sites in the North America, Europe and Japan are anticipated to recruit subjects.

1007779

#### 3.5.1. Inclusion Criteria

Refer to protocol section 4.2 for inclusion criteria.

#### 3.5.2. Exclusion Criteria

Refer to protocol section 4.3 for exclusion criteria.

# 3.6. DETERMINATION OF SAMPLE SIZE

Approximately 374 subjects will be randomized 1:1 to bexagliflozin tablets (20 mg) + sitagliptin tablets (placebo), or bexagliflozin tablets (placebo) + sitagliptin tablets (100 mg). The sample size calculation for this study was based on a two group t-test with a one-sided significance test at the 2.5% level and the following assumptions:

- 1. The non-inferiority limit (margin) for mean change from baseline to week 24 in HbA1c comparing bexagliflozin group to sitagliptin group will be 0.35%. The proposed noninferiority margin of 0.35% was based on a published clinical trial that demonstrated the effectiveness of sitagliptin, 100 mg, on HbA1c reduction in subjects with type 2 diabetes mellitus (Charbonnel, et al, 2006; Diabetes Care, 29, 2638). The sitagliptin study included male and female adult subjects with T2DM diagnosis and inadequate glycemic control defined by an HbA1c  $\geq$  7.0% and  $\leq$  10% while taking metformin monotherapy at a stable dose of ≥ 1500 mg per day. In THR-1442-C-423 study, the eligibility included the same criteria except the HbA1c range was between 7.0% to 11%. Baseline HbA1c values in the sitagliptin study was  $8.03 \pm 0.82\%$  in the placebo arm and  $7.96 \pm 0.81\%$  in the active arm, respectively. This is nearly identical to the overall baseline mean HbA1c of 7.99 ± 0.868% in the THR-1442-C-423 subject population. A placebo adjusted least-squares mean (95% CI) treatment effect of reduction from baseline in HbA1c was -0.65% (-0.77 to -0.53). The clinical meaningful margin is selected to be approximately half of sitagliptin effect, 0.35% reduction. That is, if the upper bound of 95% CI of the difference between sitagliptin and bexagliflozin is less than the chosen margin of 0.35%, the study would demonstrate that the effect of sitagliptin is preserved in the bexagliflozin treatment arm.
- 2. The pooled SD for the change from baseline to week 24 in HbA1c for bexagliflozin group and sitagliptin group will be 1.0%.

Under the above assumptions, an estimated sample size of 172 patients is needed in each treatment arm to detect non-inferiority of bexagliflozin to sitagliptin with respect to change in HbA1c at week 24 from baseline. This estimation is based on a one-sided ttest with 90% power at a 2.5% level of significance. A sample size of 187 per arm has been selected to account for approximate 8% drop-out rate and to allow adequate safety evaluation. The total sample size for this study will be 374 subjects.

1007779

#### 3.7. TREATMENT ASSIGNMENT & BLINDING

# 3.7.1. Treatment Assignment

The study will be conducted at multiple investigative sites and will involve variable numbers of subjects at each site. Enrollment will be on a competitive basis, but each site will be capped at 30 randomized subjects. Activation of investigational sites in each country will be centrally controlled by an Interactive Web Response System (IWRS).

Eligible subjects who complete the run-in period and meet all study inclusion/exclusion requirements will be randomized in a 1:1 ratio to receive active bexagliflozin with placebo sitagliptin or active sitagliptin with placebo bexagliflozin. Subjects will be assigned to treatment groups in sequential order as they qualify for the study. Randomization will be stratified according to screening (Visit V1) HbA1c (< 8.5% or  $\ge 8.5\%$ ). The investigator or designated staff will log into the IWRS to receive the randomization code and assigned kit numbers.

## 3.7.2. Blinding

This is a double-blind, double-dummy study. The sponsor, investigators, study coordinators, pharmacists, study subjects, the cardiovascular endpoint committee (CEC), and the DKA committee will be blinded to the study medications. To maintain blinding of the individual treatment assignment, the results of urinary glucose testing will not be made available to any study personnel or subjects. If knowledge of the test results is needed to manage a subject's condition, the investigator will contact the IWRS to obtain the treatment assignment. If unblinding occurs for any reason, the time and reason for breaking the blind will be recorded on the case report form (CRF) and the sponsor must be notified within 24 h. A designated statistician who is not involved with the study operation will hold the treatment codes. The unblinded treatment information can be provided to the Data and Safety Monitoring Board (DSMB) to facilitate the evaluation of any clinically important increase in the rate of a serious suspected adverse reaction or to the designated safety contact when the treatment information is required to determine if an expedited safety report must be submitted to regulatory agencies. The treatment assignment will continue to be withheld from the CEC and DKA adjudication committee members until all global investigational studies are completed and final analyses to assess cardiovascular and ketoacidosis risks are conducted.

# 3.8. ADMINISTRATION OF STUDY MEDICATION

The following investigational products will be used for oral administration:

• Bexagliflozin tablets, 20 mg: tablets containing 20 mg of bexagliflozin

1007779

• Bexagliflozin tablets, placebo: tablets containing no bexagliflozin

The following active comparator products will be used for oral administration:

- Sitagliptin tablets, 100 mg: tablets containing 100 mg of sitagliptin
- Sitagliptin tablets, placebo: tablets containing no sitagliptin

Bexagliflozin tablets, 20 mg or placebo, should be taken at approximately the same time each day, before or after breakfast, with one cup (250 mL) of water.

On the day of scheduled clinic visits when there is fasting and blood is to be drawn, administration of bexagliflozin should be delayed until after blood is drawn and taken in the clinic or at home with one cup (250 mL) of water.

Sitagliptin tablets, 100 mg or placebo, should be taken once daily at the same time as bexagliflozin, before or after breakfast, with one cup (250 mL) of water.

On the day of scheduled clinic visits when there is fasting and blood is to be drawn, administration of sitagliptin should be delayed until after blood is drawn and taken in the clinic or at home with one cup (250 mL) of water.

# 3.9. STUDY PROCEDURES AND FLOWCHART

The activities that must be performed at each clinic visit are presented in Table 1. The required laboratory tests scheduled at each visit are listed in Table 2.

A visit window of  $\pm$  3 days is allowed for all visits except Visit 3. Visit 3 is the day of randomization and the basis for the visit window.

The study staff will contact each subject prior to a scheduled clinic visit to confirm the time of the visit and to remind the subject of proper fasting practice. A subject must be queried to assess compliance with an approximately 10 hours fast prior to blood draw to ensure the FPG and triglycerides values can be accurately determined. If a subject has not fasted for approximately 10 hours, the subject must return as soon as can be arranged (within 1 week) to provide a specimen after proper fasting. Blood samples will be transported to the central lab for analysis.

Statistical Analysis Plan Theracos Sub, LLC

Version 1.0 THR-1442-C-423

**Table 1** Schedule of Events

| Procedure | Screening | Run-in | Treatment | | | | | Follow-up |
|---|---|---|---|---|---|---|---|---|
| Visit Number | V1/<br>Screening | V2/<br>Run In | V3/<br>Randomization | V4/<br>6 weeks | V5/<br>12 weeks | V6/<br>18<br>weeks | V7/ End of<br>Treatment | V8/<br>Follow up |
| Time to Randomization | -3 | -1 | 0 | 6 | 12 | 18 | 24 | 26 |
| Informed Consent | X | | | | | | | |
| Screening for I/E Criteria | X | | X | | | | | |
| Medical History | X | | | | | | | |
| Diet and Exercise Counseling | | X | | | | | | |
| Physical Examination | | | X | | | | | X |
| Abbreviated Physical Examination | X | | | | | | X | |
| Vital Signs | X | | X | X | X | X | X | X |
| Measure Weight | X | | X | X | X | X | X | X |
| Electrocardiography | X | | X | | | | X | X |
| Clinical Laboratory Tests | X | | X | X | X | X | X | X |
| Diary and Glucometer Dispensation | | X | | | | | | |
| Dispensing Run-in Drug | | X | | | | | | |
| Diary and Glucometer Record Review | | | X | X | X | X | X | X |
| Dispensing Investigational Product | | | X | | X | | | |
| Adverse Events Assessments | | X | X | X | X | X | X | X |
| Concomitant Medication Assessments | | X | X | X | X | X | X | X |

Statistical Analysis Plan Theracos Sub, LLC

Version 1.0 THR-1442-C-423

**Table 2** Schedule of Clinical Laboratory Tests

| | Screening | Run-in | Treatment | | | | | Follow-up |
|---|---|---|---|---|---|---|---|---|
| Visit number | V1/ | V2/ Run In | V3/Randomi- | V4/ | V5/ | V6/ | V7/ End of | V8/ |
| | Screening | | zation | 6 weeks | 12 weeks | 18 weeks | Treatment | Follow up |
| Time to Randomization Visit (weeks) | -3 | -1 | 0 | 6 | 12 | 18 | 24 | 26 |
| Hematology | X | | X | X | X | X | X | X |
| Serum Chemistry and Electrolytes | X | | X | X | X | X | X | X |
| Glycemic Control | X | | X | X | X | X | X | X |
| Serum Lipids | X | | X | | X | | X | X |
| Urinalysis | X | | X | X | X | X | X | X |
| Infectious Disease Testing | X | | | | | | | |
| Urine Pregnancy Test (WOCBP) | X | | X | X | X | X | X | X |

# 4. ENDPOINTS

#### 4.1. PRIMARY EFFICACY ENDPOINT

Change in HbA1c from baseline at week 24

# 4.2. SECONDARY EFFICACY ENDPOINTS

The key secondary efficacy endpoints include:

- Change in FPG from baseline at week 24
- Change in body weight in subjects with baseline BMI  $\geq$  25 kg/m<sup>2</sup> at week 24
- Change in SBP from baseline at week 24

The exploratory secondary efficacy endpoints include:

- Proportion of subjects with HbA1c of < 7% over time
- Change from baseline in HbA1c over time
- Change from baseline in FPG over time
- Change from baseline in body weight over time
- Change from baseline in SBP over time

## 4.3. SAFETY ENDPOINTS

- AEs
- AE of special interest
- Clinical laboratory results
- Physical exam results
- Vital signs
- ECG results
- Medication use

1007779

#### 5. ANALYSIS SETS

#### 5.1. SCREENED ANALYSIS SET

The Screened Analysis Set will include all subjects screened for eligibility prior to randomization. The screened population will include screen failures. Unless specified otherwise, this population will be used for summaries of subject disposition.

#### 5.2. SAFETY ANALYSIS SET

All subjects who are randomized and take at least one dose of each double-blind study medications will be included in the Safety Analysis Set. Safety analyses will be based on the medications that were taken first. The Safety Analysis Set is the primary analysis set for safety evaluation.

#### 5.3. INTENTION TO TREAT ANALYSIS SET

All subjects who are randomized regardless of treatment adherence or availability of follow up data will be included in the Intention to Treat (ITT) Analysis Set. All analyses of the ITT Analysis Set will be based on each subject's randomized assigned treatment. The ITT analysis set will serve as the primary set for the efficacy analyses.

# 5.4. PER PROTOCOL ANALYSIS SET

The Per Protocol (PP) Analysis Set will include all subjects in the ITT who meet the study eligibility requirements and have no major protocol deviations that affect the validity of the efficacy measurements. Protocol deviations that may result in subject or visit exclusion from the PP Analysis Set are described in Section 5.5. The PP analysis set will serve as the secondary set for efficacy assessment.

# 5.5. PROTOCOL DEVIATIONS

Protocol deviations will be captured during monitoring visits and recorded in CRF. Deviation will be classified into each of the 9 categories: enrollment criteria, non-compliance, laboratory, dosing, visit schedule, visit/procedure requirement, concomitant medication, informed consent, and other. Date and details of the deviation will be recorded. The list of deviation will be reviewed before unblinding and major protocol deviations that, in the opinion of the medical monitor, could affect the primary and secondary variables will be determined. Some possible types of major protocol deviations are showing in Table 3.

 Table 3
 Some Possible Types of Major Protocol Deviations

| Category | Criteria | Exclusion |
|---|---|---|
| Inclusion/Exclusion Criteria | | |
| Ineligible subject is enrolled | <ul> <li>Subjects not satisfying HbA1c inclusion criteria</li> <li>Treated with SGLT2 within 3 months of screening</li> </ul> | Subject exclusion |
| Prior or Concomitant<br>Medication Restrictions | | |
| Use of another SGLT2 inhibitor | Use of an SGLT2 inhibitor as the rescue medication for hyperglycemia | Visit exclusion [exclude data post SGLT2 starts] |
| Use of new Diuretic medication | Initiate of new diuretic medication within 12 weeks of randomization | Visit exclusion [exclude data post initiation of a new diuretic] |
| Randomization/Blinding | | |
| Unblinding | Blind was broken (requested in IWRS) | Visit exclusion [exclude data post blind broken] |
| Dosing Non-Compliance | -Subject missed more than 50% of the investigational product doses between week 12 and week 24 | Subject exclusion |

1007779

# 6. GENERAL ASPECTS FOR STATISTICAL ANALYSIS

#### 6.1. GENERAL METHODS

Statistical methodology and analyses are in accordance with the principles outlined by the International Conference on Harmonization (ICH) E9 guidelines. All statistical analyses will be conducted using SAS statistical software version 9.3 or higher.

Tables, listings and figures (TLFs) will be produced in accordance with the principles outlined by the ICH E3 guidelines. For most summary statistics, data will be analyzed by the following treatment groups: Bexagliflozin 20 mg; Sitagliptin 100 mg.

Data summaries will use descriptive statistics (number of subjects [n], mean, standard deviation [SD], 1<sup>st</sup> quartile [Q1], median, 3<sup>rd</sup> quartile [Q3], minimum and maximum) for continuous variables, and frequency and percentage of subjects for categorical and ordinal variables, unless otherwise specified.

Unless otherwise specified, all statistical tests will be one-sided using a 0.025 level of significance. All confidence intervals (CIs) will be two-sided 95% CIs.

The analysis visit window will be assigned to data collection. One selected data point per visit will appear in summary tables and figures. Refer to section 6.4 for details. All visit assessment data will be included in shift tables and will appear in the subject listings.

No data imputation will be applied for missing values, unless otherwise specified.

#### 6.2. KEY DEFINITIONS

## 6.2.1. Baseline Values

For subject who is dosed, baseline is defined as the last non-missing value on or prior to the first dose of double-blind study medication. For subject who is not dosed, baseline is defined as the last non-missing value on or prior to the randomization date.

#### 6.2.2. First Dose Date

Two "first dose dates" will be required - one for the Run-In period and one for the double-blind treatment period. The first dose date for the Run-In period will be the date of administration of the first dose of single-blind placebo tablets during the Run-In period. The first dose date for the double-blind treatment period will be the date that the first dose of randomized, double-blind study drug is administered. Both first dose dates will be obtained from the electronic case report form (eCRF). Study analyses will use the double-blind treatment period first dose date.

1007779

# **6.2.3.** Study Day

Study Day is the number of days starting from the first administration of double-blind study drug, which is counted as Study Day 1. If the assessment date is after the date of the first double-blind medication, the study day is calculated as date of assessment - date of the first dose administration+1. If the assessment date is prior to the date of the first double-blind medication, the study day is calculated as date of assessment - date of the first dose administration.

#### 6.2.4. Duration

Duration of double-blind treatment will be determined as Double-Blind duration = Double-Blind last dose date minus Double-Blind first dose date plus 1. Duration of Run-In period will be determined as Duration = last dose date in the run-in period minus first dose date in the run-in period plus 1.

# 6.2.5. End of Study

The end of study is defined as the date of final contact as entered on the End of Study page of the eCRF.

# 6.2.6. Patient Years

Patient years are calculated as sum of the duration from first dose of double-blind treatment to the end of study / 365.25 of all subjects in the specified analysis set and treatment arm. This is used as the denominator of the computation of incidence rate.

#### 6.3. MISSING DATA

The handling of missing or incomplete data is described for each endpoint and data type (as needed) in Section 7 to 9.

#### 6.4. ANALYSIS VISIT WINDOWS

Table 4 shows how data will be mapped to analysis visits prior to selection of records for analysis. All post-baseline visits, including unscheduled and early termination visits, will be mapped. After mapping the data to the analysis visits, the following rules will apply unless other handling is specified for a particular analysis.

- If multiple records are available within a single analysis visit window, the record closest to the planned assessment day will be selected for analysis.
- If 2 records are equidistant from the target day, then the later record will be selected.

1007779

• If a subject has no record in an analysis window, the subject will be considered missing at that visit.

Table 4 Analysis Visit Windows

| Study Day Window | Scheduled day | Scheduled Visit/Week |
|------------------|------------------------------|----------------------|
| Day 1 - 63 | Day 42 | Visit 4/Week 6 |
| Day 64 - 105 | Day 84 | Visit 5/Week 12 |
| Day 106 - 147 | Day 126 | Visit 6/Week 18 |
| >= Day 148 | Day 168 or (Last dose date + | Visit 7/Week 24 |
| | 1), select the less one | |

<sup>\*</sup> Week 24 is the end of treatment visit for those subjects completing the study per protocol. For endpoints of lab, vital sign and ECG, the first collection after assigned Week 24 and > 7 days from Week 24 visit will be considered as Week 26 visit. All data summary will base on the mapped visit.

#### **POOLING OF CENTERS 6.5.**

Subjects will not be pooled based on site size, but rather by region, to ensure a sufficient number of subjects per treatment arm in both ITT and PP populations for analysis that contain region as a model effect.

| Region | Country |
|------------------|---------------|
| North<br>America | United States |
| | Czech Rep |
| _ | Hungary |
| Europe | Poland |
| | Spain |
| Asia | Japan |

1007779

# 7. DEMOGRAPHIC, OTHER BASELINE CHARACTERISTICS AND MEDICATION

#### 7.1. SUBJECT DISPOSITION AND WITHDRAWALS

Subject disposition data will be listed. A disposition table will present, by treatment group and overall, the number and/or percentage of subjects who signed the informed consent and entered the study (i.e., were screened, screen failed prior to Run-in, screen failed during the Day -7 to Day -1 Run-in, and randomized), completed the study drug, discontinued study drug, completed the study, and discontinued from the study after randomization. The reasons for early withdrawal after randomization will be summarized. A separate table will display the number of subjects who met eligibility criteria at screening and Run-in period but withdrew prior to randomization (non-randomized subjects) with a summary of the reasons for withdrawal prior to randomization.

Assignment to the analysis sets (safety, ITT, and PP) will be summarized.

#### 7.2. SUBJECT ELIGIBLITY AND PROTOCOL DEVIATIONS

All subjects, including screen failure subjects, who violate the Inclusion/exclusion criteria will be listed. Reason for screen failure will be summarized.

Deviations that could affect the primary and secondary variables will be considered when determining a subject's eligibility for the PP population. The number and percent of subjects who had any major deviation and each type of major protocol deviation will be tabulated for the ITT Analysis Set.

#### 7.3. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Demographic characteristics include age, gender, race and ethnicity. Subject age will be calculated from the date of informed consent date. Baseline characteristics will include HbA1c, baseline HbA1c group ( $\leq 8.5\%$  vs. > 8.5%) at Visit 1, blood pressure, body weight, BMI, FPG, eGFR, duration of diabetes from diagnosis to the date of informed consent, and prior anti-diabetic treatment status at screening (including type of therapy used, such as metformin, SU, DPP-4 inhibitor, alpha-glucosidase inhibitor, etc.). Descriptive summary statistics by treatment will include counts and percentages for discrete variables and estimation of means, standard deviations, medians, inter-quartile range (Q1, Q3), minimum, and maximum for continuous variables. Subjects' baseline demographic and baseline characteristics will be summarized by treatment group and overall for subjects in the safety, ITT, and PP analysis set.

1007779

#### 7.4. MEDICAL HISTORY

Significant medical and surgical history, including dates of diagnoses and procedures and whether the condition is ongoing, if applicable, will be collected. Each condition will be recorded as a verbatim term, date of onset, date resolved, and a checkbox that indicates ongoing conditions. Significant surgical and medical history will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 19.0.

Medical and surgical history will be summarized for the Safety Analysis Set by treatment group, system organ class (SOC), and MedDRA preferred term (PT), overall. Subject data will be listed.

Subject diabetes and cardiovascular diseases history will be summarized for all categorical variables by frequency and percentage. Listing will be provided.

#### 7.5. MEDICATION

All prescription and over-the-counter medications, including vitamins and herbal supplements, that subjects receive during the trial must be documented on the CRF. The medication name, dose, frequency, route of administration, date(s) of administration and reason for administration must be recorded. This documentation should continue through the treatment period and the follow up period.

All medication will be coded using the World Health Organization Drug Dictionary (WHO-DD) version March 2016. Preferred drug name, Anatomical Therapeutic Chemical (ATC) class will be reported for inclusion in the database.

Medication summaries based on ATC level 2, and the preferred drug names will be produced for the Safety Analysis Set. The summaries will present, by treatment group, the frequency and percentage of subjects who used any medication in an ATC class, or any medication based on a single preferred drug name. Medication summaries will be sorted by descending total frequency of ATC class and by PT within ATC class. Subjects will be counted only once for each medication class and each preferred drug name.

For subject listings, ATC class and PT of the medications will be reported; multiple medications for an individual subject will be listed by start date and then by stop date, from earliest to latest medications.

# 7.5.1. Prior Medication

Any medication stopped prior to the first dose of the double-blind treatment period will be considered a prior medication.

1007779

No summary for prior medication will be presented. Prior and concomitant medications will be presented together on a single listing. Prior medication will be indicated in the listing.

#### 7.5.2. Concomitant Medication

A concomitant medication is any medication that the subject has been taking prior to the first dose of double-blind study medication and that the subject is expected to continue to take for some portion of the study treatment period, as well as any medication other than the investigational product that the subject takes during the double-blind treatment period and follow up period of the study. In the case of completely missing stop date, medication will be assumed to be concomitant. If a medication can be considered as both prior and concomitant due to partial stop date, it will be considered as concomitant.

Any medication a subject takes to treat hyperglycemia after the first dose of double-blind study drug starts and continues for more than 2 weeks before study treatment stops is considered a rescue therapy and should be recorded in the concomitant medication log. Increase total daily dose of metformin, the background hypoglycemic therapy, is also considered rescue medication if the dose is intensified during the double-blind treatment period for more than 2 weeks before study treatment stops. All medication given to treat hyperglycemia will be recorded in CRF.

Concomitant medications will be presented in a summary table as well as in a subject listing. Rescue medications will be summarized in a separate table and will be indicated in the same listing.

1007779

#### 8. EFFICACY

Efficacy data include HbA1c, FPG, body weight, and SBP. For subject who is dosed, changes from baseline will be calculated as the post-treatment value minus the last non-missing value on or prior to the first dose of double-blind study medication. For subject who is not dosed, changes from baseline will be calculated as the post-treatment value minus the last non-missing value on or prior to the randomization date. All continuous efficacy data will be summarized for observed and change values by treatment and visit. Proportion of subjects with HbA1c of < 7% will be summarized by frequency and proportion by treatment and visit.

# 8.1. PRIMARY EFFICACY ENDPOINT AND ANALYSIS

The primary efficacy hypothesis is that bexagliflozin reduces HbA1c after 24 weeks of treatment when compared to sitagliptin.

# 8.1.1. Primary Efficacy Analysis

Let  $\mu_{Bexagliflozon}$  and  $\mu_{sitagliptin}$  represent the mean changes from baseline in HbA1c at Week 24 for bexagliflozin and sitagliptin arms, respectively. The following hypotheses will be tested:

H0:  $\mu$  bexagliflozin -  $\mu$  sitagliptin >  $\delta$  Ha:  $\mu$  bexagliflozin -  $\mu$  sitagliptin  $\leq \delta$ 

This hypothesis will be tested based on ITT analysis set using all observed data and a mixed model repeated measures (MMRM) approach. The MMRM model will include treatment, visit, treatment-by-visit interaction, region and the baseline HbA1c value as a fixed effect covariate. The analysis will evaluate the mean change from baseline in HbA1c over the 24-week double-blind treatment period. An unstructured covariance will be used to model the within-subject correlation. The Kenward-Roger approximation will be used to estimate denominator degrees of freedom. If the model with the unstructured covariance structure does not converge, an autoregressive(1) covariance structure will be used. HbA1c values obtained after the start of rescue medication will not be excluded from the analysis.

Based on the MMRM model, the treatment and treatment-by-visit interaction terms allow for comparisons of the treatment groups at each visit, and over week 6 to week 24. Least squares (LS) mean treatment differences between the bexagliflozin group and the sitagliptin group at week 24 will be estimated from the model with their two-sided 95 % CIs presented.

Descriptive statistics (n, mean, Q1, median, Q3, SD, minimum, and maximum) will be reported by treatment group and visit, along with the LS means, differences between LS

1007779

means, a 2-sided 95% confidence interval for each difference from the model effects. In addition, the LS means with standard errors (SEs) of the change from baseline over time and difference between treatment groups with 95% CIs will be presented graphically for the ITT population.

In non-inferiority analysis, a CI is calculated to estimate the range of values in which the treatment difference is likely to lie. This CI is used to provide the basis for drawing the study's conclusions. In this specific test, if the 95% CI lies below the specified non-inferiority margin 0.35%, the results would lead to a conclusion of non-inferiority of bexagliflozin treatment to sitagliptin treatment. Superiority of bexagliflozin group over sitagliptin group at week 24 in HbA1c change from baseline will be declared if the upper bound of 95% CI is less than 0.

For supportive analyses, the primary efficacy endpoint will be analyzed with observed available data using the PP analysis set in a similar manner as above.

# 8.1.2. Sensitivity Analyses

Randomized subjects who withdraw consent to participate in the study will not be replaced. The early termination rate is estimated to be 8%. To the extent possible, attempts will be made to minimize the amount of missing data through measures planned in the study conduct.

To investigate the possible implications of missing values in efficacy assessments, the number, timing, pattern, and reason for the missing value will be summarized. The reason for withdrawn will be reviewed. If there are missing values for the primary analysis, only available data will be analyzed and data obtained after rescue will not be excluded. To account for subjects for whom the post-baseline endpoint (ie, at the time when the last post-baseline double-blind assessment was performed) occurs at a time point before Week 24, a MMRM approach will be used as the primary method (as described in the previous section). It is assumed that the majority of the missing values will be one of the following, and in such situations, likelihood-base methods like MMRM are appropriate and widely accepted (Little et al, 2002):

- "Missing Completely at Random (MCAR)" (ie, probability of an observation being missing does not depend on observed or unobserved measurements) or
- "Missing at Random (MAR)" (ie, probability of an observation being missing depends only on observed measurements)

The dropout patterns will be assessed by a Kaplan-Meier plot of time to discontinuation by treatment group to assess whether they differ between treatment groups.

1007779

The following sensitivity analyses will be conducted:

- 1) Missing data will be imputed via multiple imputations, following which the MMRM will be repeated on the complete datasets with results combined across complete datasets using standard multiple imputations techniques; HbA1c values collected after the start of rescue medication will not be excluded. A pattern-mixture model will be used to explore the impact of the missing data. Imputation will be conducted within each treatment arm and subgroup (treatment completer vs. treatment terminated early) under the assumption that non-adherent subjects with missing data will follow the same trajectory of non-adherent subjects with values observed. All efforts will be made to retain subjects in the study. If treatment is discontinued, subjects are encouraged to remain in the study and complete all scheduled visits, including final follow-up visit. However, with all efforts, insufficient values may be available for reliable imputation. This analysis will be performed only if ≥3% of subjects in each treatment arm completed scheduled week 24 visit after treatment is stopped. For this analysis, the following three-step approach outlined below will be used:
  - a. Non-monotone (intermediate visits) missing data will be imputed first using the Monte Carlo Markov Chain (MCMC) method under the MAR assumption in all treatment arms (using the MCMC statement in PROC MI). Multiple chains option (CHAIN=MULTIPLE option in the MCMC statement of PROC MI) will be used. For the non-monotone imputation of the HbA1c missing data, a multivariate normal model will be used including variables for the HbA1c at baseline and all post-baseline visits within each treatment group.
  - b. After the non-monotone missing data have been imputed, the remaining monotone missing data will be imputed within each treatment arm and subgroup, defined by whether subject completed 24 week of study treatment, using regression approach. The predictors for the regression imputation model at any time point will be region, and HbA1c at all previous time points, including baseline. Imputations will be performed using a sequence of regression-based imputations (using PROC MI statement MONOTONE REG) at each post-baseline time point.
  - c. Imputed data in each of the multiple imputed datasets will be analyzed using the same mixed model for repeated measures as in the primary analysis. The results from all imputed datasets will be combined using the Rubin's combination rule (PROC MIANALYZE).

The number of imputation will be determined using the method described by White, et.al., 2011. We will use Bodner's approximation to estimate the fraction of missing information (FMI) as the proportion of the incomplete cases in the data. Since the parameter of interest is the mean changes from baseline in HbA1c at Week 24 for bexagliflozin and sitagliptin groups, FMI will be approximated using the

1007779

proportion of subjects missing Week 24 values. As indicated by Bodner, this is a very conservative approach and will work with FMI≤0.5. The number of imputations m will be determined to provide sufficient level of reproducibility using formula:

m≥100×FMI

as recommended by White. The Monte Carlo error of the p-value using m imputation datasets will be approximately 0.01 when the true p-value is 0.05, and 0.02 when the true p-value is 0.1.

At least 10 datasets will be imputed. We will examine the FMI estimated from the combined results. If it is much larger than our initial approximation, a considerable volatility is observed from the imputed datasets. In this case, we will increase the number of m using the estimated FMI.

- 2) Additionally, the impact of the data after the start of rescue medication will be evaluated. HbA1c values collected after the start of rescue medication will be considered missing, and the MMRM analyses will be performed. Same statistics provided for the primary analysis will be presented.
- 3) Tipping point analysis will be conducted. Data after rescue medication will be considered as missing. Following steps will be followed:
  - a. Create monotone missing data as step a in 1);
  - b. Regression approach under MAR will be used to generate complete datasets. The predictors for the regression imputation model at any time point will be region, treatment, and HbA1c at all previous time points, including baseline. The first imputed values will be penalized or rewarded based on the treatment subject received:
    - o Subjects in the bexagliflozin group: missing value will be analyzed assuming the treatment effect is worsened by  $\delta 1$  (where  $\delta = 0.1$  to 0.5, in step of 0.1) compared to the subjects who have no missing value in the reduction of HbA1c value;
    - $\circ$  Subjects in the sitagliptin group: missing value will be analyzed assuming the treatment effect is better by  $\delta 2$  (where  $\delta = 0.1$  to 0.5, in step of 0.1) compared to the subjects who have no missing value in the reduction of HbA1c value;

The penalty or reward will not be applied to the values from later time points as these values are penalized or rewarded through regression on previous time points.

1007779

c. Imputed datasets will be analyzed and results combined as step c in 1).

For each combination of  $(\delta 1, \delta 2)$ , 100 imputed datasets will be obtained. These 25 combinations will be separately analyzed to explore under which condition when the null hypothesis can no longer having evidence to be rejected.

#### 8.1.3. Subgroups

The primary efficacy endpoint will be summarized and analyzed by the following subgroups using MMRM model:

- Age (<65 years or ≥65 years), adjusted by region and baseline HbA1c value;
- Gender (male or female), adjusted by region and baseline HbA1c value;
- Race (Asian; Black of African American; White or Caucasian; Other), adjusted by region and baseline HbA1c value;
- Baseline HbA1c (>8.5% or  $\leq$  8.5%), adjusted by region;
- Region (North America, or Europe, or Asia Pacific), adjusted by baseline HbA1c value.

#### 8.2. SECONDARY EFFICACY ENDPOINT(S) AND ANALYSES

The secondary endpoints will only be tested when the non-inferiority of the primary efficacy assessment is established at one-sided significance level of 0.025. To control the overall type I error of 0.025 one-sided, the secondary efficacy objectives will be tested at one-sided 0.025 significance level following the hierarchy sequence as below:

- Superiority test of the change in FPG in the bexagliflozin group vs. the sitagliptin group at week 24.
- Superiority test of the change in body weight in subjects with baseline body mass index (BMI)  $\geq$  25 kg/m<sup>2</sup> in the bexagliflozin group vs. the sitagliptin group at week 24.
- Superiority test of the change in SBP in the bexagliflozin group vs. the sitagliptin group at week 24.

Analysis for secondary endpoints will be based on ITT analysis set and repeated for PP analysis set.

#### 8.2.1. Change in FPG in the bexagliflozin group vs. the sitagliptin group at week 24

This will be tested if the non-inferiority of HbA1c has been concluded based on ITT

1007779

analysis set. Data after rescue medication will not be excluded. The comparison of change in FPG between randomized treatments at week 24 will be carried out using the similar MMRM model as in section 8.1.1. The model will include terms for treatment, visit, treatment-by-visit interaction, region as fixed effects and the corresponding baseline FPG value as covariate. Treatment comparison p-values and difference at week 24 will be estimated from the model, with the two-sided 95 % CIs of the treatment difference also presented. If the inferiority of HbA1c is not established, the nominal p-value will not be used for inferential purposes. Summary table will be presented and figures will be displayed for ITT analysis set.

# 8.2.2. Change in body weight in subjects with baseline body mass index (BMI) ≥ 25 kg/m² in the bexagliflozin group vs. the sitagliptin group at week 24

This will be tested if the non-inferiority of HbA1c has been concluded and the previous secondary efficacy endpoint of FPG reduction is in favor of bexagliflozin significantly. Change from baseline in body weight at week 24 will be analyzed in a similar manner as change in FPG, Section 8.2.1, based on ITT analysis set for all subjects. Baseline body weight will be used as a covariate. Region and baseline HbA1c value will also be used as fixed effects. Summary table will be presented and figures will be displayed for ITT analysis set.

# 8.2.3. Change in SBP in the bexagliflozin group vs. the sitagliptin group at week 24

This will be tested if the non-inferiority of HbA1c has been concluded and the previous secondary efficacy endpoints (reduction in FPG and body weight) are significant in favor of bexagliflozin. Change from baseline in SBP at week 24 will be analyzed in a similar manner as change in FPG, Section 8.2.1, based on ITT analysis set for all subjects. Baseline SBP will be used as a covariate. Region and baseline HbA1c value will also be used as fixed effects. Summary table will be presented and figures will be displayed for ITT analysis set.

# 8.2.4. Sensitivity analysis

For all secondary analyses of FPG, body weight and SBP, missing data will be imputed via multiple imputations, following which the MMRM will be repeated on the complete datasets with results combined across complete datasets using standard multiple imputations techniques; Values collected after the start of rescue medication will be considered missing. Imputation steps include:

- a. Create monotone missing data as step a in 1) of section 8.1.2;
- b. Regression approach under MAR will be used to generate complete datasets. The

predictors for the regression imputation model at any time point will be region, treatment, and values at all previous time points, including baseline. Values at each visit will be imputed sequentially. The first imputed values for subjects in bexagliflozin arm will be penalized by the mean improvement at week 24 on that endpoint (i.e. the mean change from baseline at week 24). Imputed values for subjects in sitaglipin will not be penalized. Imputed values after the first missing value will be penalized through regression on first penalized value.

c. Imputed datasets will be analyzed and results combined as in step c in 1) in section 8.1.2.

#### 8.3. EXPLORATORY EFFICACY ENDPOINTS AND ANALYSES

All endpoints in this section are exploratory. No sensitivity analysis and adjustment for multiple comparisons will be conducted. Nominal p-values will be used to examine any trends in these endpoints.

# 8.3.1. Change from baseline in HbA1c, SBP, Body weight, and in FPG over time

The schedule of HbA1c, FPG, body weight, and SBP/DBP can be found in Table 1. The absolute value and change from baseline in HbA1c, FPG, body weight and SBP during the double-blind treatment period will be summarized by descriptive statistics at each visit. Change from baseline in HbA1c will be analyzed as part of primary efficacy analysis (Section 8.1.1). Change from baseline in SBP, body weight and FPG will be analyzed as part of key secondary analysis (Section 8.2.1, 8.2.2, and 8.2.3). LS means for each treatment and the difference between treatments will be estimated at each visit. The corresponding p-values will also be presented.

All values for follow-up visits will be listed.

# 8.3.2. Proportions of subjects with HbA1c of < 7% over time

Summary on the proportion of subjects achieving HbA1c < 7% at each visit will be presented over time. It will be analyzed using Generalized Estimating Equation (GEE) logistic regression. The fixed effect will include region, treatment, visit, treatment-by-visit interaction and baseline HbA1c. An unstructured correlation structure will be used (or autoregressive (1) if the model with the unstructured structure does not converge). The odds ratios of bexagliflozin group over the sitagliptin group at each visit will be estimated from LS means based on the model with the corresponding p-values and their two-sided 95 % CIs presented.

1007779

#### 9. SAFETY

The analysis population used for safety analyses will be the Safety Analysis Set. Safety data include AEs; physical examination results; vital signs, including blood pressures; ECG results; and clinical laboratory results, including serum chemistry, hematology, serum lipids, and urinalysis.

Observed data will be summarized by treatment group as counts and percentages for discrete variables and means, standard deviations, medians, inter-quartile range, minimum, and maximum for continuous variables. All subjects who are randomized and receive at least one dose of double-blind study medication will be included in the safety analysis. All safety data will be presented in by-subject listings and included in the clinical trial report.

#### 9.1. EXTENT OF EXPOSURE

Study drug exposure will include:

- Treatment duration by treatment group
- Total dose received by treatment group

Treatment duration of tablets (in weeks) is calculated as (the date of the last dose of study drug - the date of the first dose of study drug + 1) / 7 and rounded to 1 decimal place.

The specific definitions of the first dose and last dose dates of study drug are given below:

- First dose date: The date of the first dose of study treatment during the double-blind treatment period obtained from the study drug exposure CRF.
- Last dose date: The date of the last dose of study medication in the 24 week treatment period for subjects who have completed the study or discontinued early. Total dose received will be calculated as number of tablets dispensed number of tablets returned.

Summary statistics for treatment duration (in weeks) and total dose received, as well as a frequency summary of treatment duration categories (e.g., < 1, 1 - < 6 weeks), will be provided.

1007779

#### 9.2. TREATMENT COMPLIANCE

Subjects will be provided with dosing instructions each time study medication is dispensed. Subjects will also be instructed to bring their medication with them to every visit. During the run-in period, subjects will be considered compliant in investigational product administration by missing no more than one day of run-in medication. Subjects who are not compliant during the run-in period will be excluded from randomization. If, in the judgment of the investigator, it was appropriate for the subject to omit these doses, this requirement may be waived (e.g., if the subject was hospitalized overnight during run-in).

At each visit after the start of the run-in period, the study staff will review the self-monitored blood glucose (SMBG) control diary and medication use with the subject and record the drug consumption in the CRF. Reasons for non-adherence will also be recorded in the protocol deviation log if applicable.

Compliance in the run-in and double-blind phase is calculated for as follows:

- Percent compliance = (number of tablets taken / number of tablets should have taken) x 100.
- Number of tablets taken = number of tablets dispensed number of tablets returned.
- Number of tablets should have taken = (number of tablets supposed to take in a day) x (number of exposure days).
- Number of exposure days = last dose date first dose date + 1.

If any of the bottles dispensed is not returned, it will not be possible to compute the compliance. In this case, the number of tablets taken and compliance will be considered as missing. Summary statistics for tablet compliance (%) will be provided by treatment group for the double-blind treatment period. A frequency summary of compliance will also be presented with the following categories: < 75%, 75-<100%, 100-120%, and > 120%.

## 9.3. ADVERSE EVENTS

Adverse events will be collected and recorded from the time a subject signs the Informed Consent Form (ICF) to the last scheduled contact. And new SAEs reported by the subject to the investigator that occur after the last scheduled contact, and are determined by the investigator to be reasonably associated with the use of the investigational product, should be reported to the sponsor or designated personnel. This may include SAEs that are captured on follow-up telephone contact or at any other time point after the defined study period (i.e., up to last scheduled contact). The investigator should follow SAEs identified after the last scheduled contact until the events are resolved, or the subject is lost to follow-up. The investigator should continue
1007779

to report any significant follow-up information to the sponsor until the event has been resolved. This study requires that subjects be actively monitored for SAEs for at least 4 weeks after the last treatment.

For all AEs, preferred AE terms and system organ class SOC will be coded using terminology from the MedDRA, version 19.0.

A Treatment-emergent Adverse Event (TEAE) is defined as an AE that begin after the first administration of double-blind study medication or existing AEs that worsen after the first dose of double-blind study medication. All reported AEs will be listed, but only TEAEs will be summarized in tables.

Drug-related AEs will be considered those to be possibly, probably and definitely related to study medication administration based on the investigators assessment.

Unless otherwise specified, AEs will be summarized by SOC and PT, with SOCs and PTs within SOCs presented in descending order of subject incidence.

#### 9.3.1. Derived Data

AE onset day is calculated as (date of AE start - date of double-blind first dose + 1) if it is after the first dose of study drug. AE onset day is calculated as (date of AE start - date of double-blind first dose) if it is before the first dose of study drug. The onset day will be missing if the start date is missing.

## 9.3.2. Data Summarization

AE summary tables are listed below:

- An overall summary of the number and percentage of subjects reporting any TEAEs, serious TEAEs, treatment-related TEAEs, serious treatment-related TEAE, any TEAEs leading to treatment discontinuation, any TEAEs leading to subject discontinuation and TEAEs leading to death.
- TEAEs overall and by SOC and PT
- TEAEs by severity, overall and by SOC and PT
- Serious TEAEs, overall and by system organ class and preferred term
- TEAEs by relationship to study treatment, overall and by system organ class and preferred term
- TEAEs leading to treatment discontinuation, overall and by SOC and PT
- TEAEs leading to study discontinuation, overall and by SOC and PT

1007779

Most common TEAEs. Most common TEAEs are defined as TEAEs that occur in
 5% of the subjects in either of the treatment groups.

For summary tables, subjects having more than 1 event with the same PT will be counted once for that term. Subjects having more than 1 event with the same SOC will be counted once for each event and once for that SOC. For tabulations by severity, only a subject's most severe event within the category (e.g. overall, SOC, PT) will be counted; similarly, for tabulations by relationship, only a subject's most related event within a category will be counted. The denominator for percentages will be the number of subjects in the Safety Analysis Set for the given treatment group (i.e., the N's for the columns).

Listings will be provided for all AEs and the following subsets:

- All TEAEs
- All TEAEs at least possibly related to study medication
- Serious AEs
- AEs leading to treatment discontinuation
- AEs leading to death

# 9.3.3. AE of Special Interest

AE of special interest includes UTI, GMI, diuretic effects, hypotension episodes, hypoglycemia, hepatotoxicity, MACE, falls and fractures, malignancy, hypersensitivity reactions, pancreatitis, amputations and renal failure events. These AEs of interest except DKA, MACE and amputations will be prospectively identified based on the MedDRA preferred terms in the AE log by a medical expert prior to the data base lock and unblinding of the individual subject treatment assignment. The list of AE of interest will be confirmed in a peer review process. DKA and MACE will be identified by the investigator and documented in the CRF, and subsequently adjudicated by separate independent committees. Adjudicated results will be used for summary. Amputation events will be recorded in the procedures and amputation CRF. Cardiovascular events, hypoglycemia events by severity, and amputations will be summarized separately.

# 9.3.3.1. AE of special interest identified by PTs

Cardiovascular events considered as MACE by investigator will be submitted to an independent CEC for adjudication. The events of interest include cardiovascular mortality, MI, stroke, hospitalization for acute coronary syndromes, urgent revascularization procedures, and other possible serious cardiovascular events. Other AE of special interest will be identified from the PTs. The number and percentage of subjects experiencing these TEAEs of special interest will be summarized for each treatment group by type of event. The incidence rate of AE of special interest per 100 patient years will also be summarized. Each category of events will be displayed in a

1007779

separate listing.

## 9.3.3.2. Hypoglycemic Events

Hypoglycemic event categories include:

| Category | Description |
|---|---|
| Severe | Assistance required and blood glucose ≤70 mg/dL or no value |
| | available but responded to glucose treatment |
| Documented | Blood glucose ≤70 mg/dL and typical symptoms of hypoglycemia |
| Symptomatic | |
| Asymptomatic | Blood glucose ≤70 mg/dL and no typical symptoms of hypoglycemia |
| Probable | Typical symptoms of hypoglycemia and no value available but |
| Symptomatic | responded to glucose treatment |
| Relative | Typical symptoms of hypoglycemia and blood glucose >70 mg/dL |

While each event meeting the criteria above will be entered into the hypoglycemia log, only critical (severe) hypoglycemia, documented symptomatic hypoglycemia, asymptomatic hypoglycemia, and probable hypoglycemia will be entered as AEs.

The number and percentage will be summarized by treatment for:

- Each category of hypoglycemic events;
- Any severe or documented hypoglycemic events.

## 9.3.3.3. Major Adverse Cardiovascular Events

Cardiovascular events considered as MACE by investigator will be submitted to an independent CEC for adjudication. The events of interest include cardiovascular mortality, MI, stroke, hospitalization for acute coronary syndromes, urgent revascularization procedures, and other possible serious cardiovascular events. The number, percentage and incidence rate per 100 patient years of suspected MACE and adjudicated MACE will be summarized for each treatment group. Adjudicated MACE will be further summarized by PTs.

## 9.3.3.4. Revascularization and Amputations

Revascularization and amputations information are collected in a separate form. Frequency and percentage will be summarized for:

- Type of procedures -cardiovascular related or amputation
- Subjects with any amputation
- Conditions that resulted in amputation

1007779

Location of amputation

Only procedures performed after the first dose of double-blind study drug will be summarized.

#### 9.4. LABORATORY EVALUATIONS

Laboratory tests will include hematology panel, chemistry panel, serum lipids, and urinalysis testing. Hematology, chemistry, and urinalysis will be performed at the following time points: at the screening visit, on randomization visit, and at week 6, 12, 18, 24, and 26. Serum lipids will be performed at the screening visit, on randomization visit, and on week 12 and 24, and 26. The study staff will contact each subject prior to a scheduled clinic visit to confirm the time of the visit and to remind the subject of proper fasting practice. A subject must be queried to assess compliance with an approximately 10-hour fast prior to blood draw to ensure the FPG and triglycerides values can be accurately determined. If a subject has not fasted for approximately 10 hours, the subject must return as soon as can be arranged (within 1 week) to provide a specimen after proper fasting. A list of laboratory tests is included in Table 5.

Low density lipoprotein cholesterol (LDL-C) will be calculated by the Friedewald equation. If triglycerides are > 400 mg/dL, the calculated LDL-C value is invalid by this equation and will be set as missing. Direct LDL-C will be determined in subjects whose triglycerides are > 350 mg/dL at screening visit. All subsequent LDL-C of these subjects will be determined by the same direct LDL-C measurements only. If triglycerides are > 350 mg/dL, a reflex test will be performed based on direct LDL measurement. The following algorithm will be used to obtain LDL-C values for the analyses:

- 1. Select subjects (based on the SI unit) who had screening triglycerides >3.4 or >350 based on the conventional unit
- 2. Take the LDL direct measurement values only, throughout the study visits for those subjects
- 3. If screening triglycerides > 350 and no direct LDL-C values have been determined, take the calculated.

Among those subjects who have screening triglycerides >350 and have both calculated and direct LDL values, only take the direct LDL.

Urinalysis microscopy will be conducted if the subject has a positive result on the leukocyte esterase or nitrite dipstick tests to clarify the significance of the finding. Results of glucose measurement in the urinalysis must be suppressed from the laboratory reports so the sponsor, investigators, study coordinators, pharmacists, study subjects, and the CEC members will remain blinded to the dosing assignment.

All continues variables will be summarized by number of subjects [n], mean, SD, Q1,

1007779

median, Q3, minimum and maximum and categorical variables will be summarized by frequency and percentage.

All scheduled and unscheduled results will be considered in tables that assess maximum grade or toxicity.

Observed values (in SI units) and change from baseline over time will be summarized by treatment group. Laboratory data will be classified as low, normal, or high relative to the parameter's reference range. Laboratory abnormalities for each treatment will also be summarized with shift tables for selected parameters.

All laboratory data will be listed. For hematology, chemistry, and serum lipids, columns will be included for normal ranges and individual abnormal laboratory values will be flagged and clinical significance will be indicated. A listing for the microscopic examination will be provided for subjects who have a positive result from the urinalysis dipstick evaluation.

1007779

**Table 5** List of Laboratory Tests

| TEST NAME | SHIPMENT |
|---|---|
| Hematology | Ambient |
| Hematocrit (Hct) | <ul> <li>Mean corpuscular volume (MCV)</li> </ul> |
| Hemoglobin (Hgb) | <ul> <li>Red cell distribution width (RDW)</li> </ul> |
| Mean corpuscular hemoglobin (MCH) | <ul> <li>Red blood cell (RBC) count</li> </ul> |
| Mean corpuscular hemoglobin<br>concentration (MCHC) | White blood cell (WBC) count with differential |
| Platelet count | |
| Serum Chemistry and Electrolytes | Ambient |
| Albumin (ALB) | Total protein |
| Alanine aminotransferase (ALT) | • Calcium (Ca) |
| Alkaline Phosphatase (ALP) | Magnesium |
| Aspartate aminotransferase (AST) | • Phosphorus |
| Blood urea nitrogen (BUN) | • Potassium (K) |
| Glucose | • Sodium (Na) |
| Bicarbonate (HCO3) | Total bilirubin |
| Creatinine | Direct bilirubin |
| Chloride (Cl) | • Uric acid |
| Glycemic Control | Ambient |
| • Fasting plasma glucose (FPG) | |
| Hemoglobin A1c (HbA1c) | |
| Serum Lipids | Ambient |
| • Total cholesterol (TC) | <ul> <li>Low-density lipoprotein cholesterol (LDL-C),</li> </ul> |
| High-density lipoprotein cholesterol | calculated |
| (HDL-C) • Triglycerides (TG) | • LDL-C, direct |
| Urinalysis | Ambient |
| Appearance | • Nitrite |
| Bilirubin | <ul> <li>Occult blood</li> </ul> |
| • Color | • pH • Protein |
| • Glucose | <ul> <li>Specific gravity</li> </ul> |
| • Ketones | Urobilinogen |
| Microscopic examination of sediment UACR | • Leukocyte esterase |
| Urine Pregnancy Test (WOCBP) | Local |

1007779

#### 9.5. VITAL SIGNS

Vital signs will be measured at the screening visit, on randomization visit, and at week 6, 12, 18, 24, and 26. Measurements of vital signs will include measurement of supine, sitting and standing BP measurements, and heart rate. Only the BP measured in the sitting position will be used to determine eligibility. Orthostatic systolic and diastolic BP will be calculated as supine measurement - standing measurement.

For BP and heart rate, observed values and change from baseline will be summarized by treatment group and mapped visit using descriptive statistics (n, mean and median, standard deviation, Q1, and Q3, minimum and maximum). For BP, supine, sitting, standing, and orthostatic BP will be summarized. Subjects vital sign measurements, including scheduled and unscheduled visits, will be listed.

#### 9.6. ELECTROCARDIOGRAM

A 12-lead ECG will be conducted at the screening visit, on randomization visit, at week 24, and at week 26. ECG parameters measured will be the RR interval, PR interval, QRS duration, and QT interval. Each ECG should also be assessed by the investigator for signs of ischemia, clinically significant hypertrophy, and clinically significant T-wave abnormalities or arrhythmia.

For each abnormal ECG result, the investigator shall ascertain if the observation represents a clinically significant change from the screening ECG for that individual subject (this determination, however, does not necessarily need to be made the first time an abnormal result is observed. The investigator may repeat the ECG to verify the results of the original result). If the ECG result is determined to be a clinically significant and abnormal change from baseline for that subject, it is considered an AE.

For the ECG parameters, observed values and change from baseline from scheduled visits will be summarized with descriptive statistics by treatment group and overall at each visit. The maximum change from baseline from scheduled visits will also be provided for ECG parameters.

For the ECG overall assessment, the number and percentage of subjects in each overall assessment category (normal, abnormal but not clinically significant, abnormal and clinically significant, missing) will be presented by treatment group and overall at each visit.

#### 9.7. PHYSICAL EXAMINATION

A complete physical examination will be conducted at the randomization visit and at week 26. The examination will include measurement of body weight, and a general assessment of all body systems including the skin, head, eyes, ears, nose, throat, neck,

1007779

heart, lungs, abdomen, lymph nodes, and extremities. An abbreviated physical examination will be conducted at screening visit and at week 24, or clinically indicated. The examination will include body weight and height (height will be measured only at screening), and general assessment of the skin, heart, lungs and abdomen. Physical examination findings will be presented in a by-subject listing.

1007779

#### 10. INTERIM ANALYSES

No interim analyses are planned.

## 11. DATA AND SAFETY MONITORING BOARD

An independent DSMB will review descriptive summaries of accumulating safety, subject disposition and limited efficacy data every 6 months, or a frequency recommended by the DSMB.

A designated statistician who is not involved with the study operation will hold the treatment codes. The unblinded treatment information can be provided to the DSMB to facilitate the evaluation of any clinically important increase in the rate of a serious suspected adverse reaction or to the designated safety contact when the treatment information is required to determine if an expedited safety report must be submitted to regulatory agencies. The data outputs for this review will be created by an unblinded team. Personnel involved in the conduct of the study will not participate in the preparation of these outputs, receive the data, or participate in the unblinded portions of the DSMB meetings. More details will be provided for DSMB charter and DSMB SAP.

#### 12. CHANGE FROM ANALYSIS PLANNED IN PROTOCOL

Protocol section 9.3.2 states "Safety analyses will be based on the medication that was actually taken by each subject." SAP is changed to use 'Safety analyses will be based on the medication that was taken first.' in section 5.2.

Protocol section 9.5.2 includes sensitivity analysis using LOCF. This has been removed after tipping point analysis is added, as LOCF is redundant.

Protocol section 9.7 states 'Cumulative summary on the proportion of subjects achieving HbA1c < 7% will be presented over time'. SAP is changed to summarize the proportion of subjects achieving HbA1c < 7% at each visit in section 8.3.2.

1007779

## 13. REFERENCE LIST

Little, R., Yau, L. Intent-to-Treat Analysis for Longitudinal Studies with Drop-Outs. Biometrics, 1996; 52: 1324–1333.

Ratitch, B., O'Kelly, M. Implementation of Pattern-Mixture Models using Standard SAS/STAT Procedures. Pharmasug 2011 - Paper SP04, PHARMASUG.

Bodner TE. What improves with increased missing data imputations? Structural Equation Modeling: A Multidisciplinary Journal 2008; 15: 651–675.

White IR., Royston P., Wood AM. Multiple imputation using chained equations: Issues and guidance for practice. Statistics in Medicine 2011; 30: 377—399.

1007779

## 14. PROGRAMMING CONSIDERATIONS

The following conventions will hold for programming of outputs:

- SAS® Version 9.4 will be used for programming and production
- The format of the table shells will be followed as closely as possible; however, in the course of programming and familiarization with the database, some changes may become necessary. All changes will be documented. Major changes will be documented through a formal amendment to this document.
- Patients in this study will be identified as "Subjects."
- Descriptive statistics will be displayed in the following order:

n Mean Standard deviation (SD) Q1, Q3 Median Minimum, Maximum

- Decimal places: For summary statistics, the minimum and maximum will be reported with the same number of decimal places as the collected measure, the mean, LS mean (if applicable) and median will have 1 more decimal place than the measure collected, and the SD and confidence interval (CI) will have 2 more decimal places than the collected measure. For frequency distributions, percentages will be reported to 1 decimal place. For p-values, 4 decimal places will be reported or the SAS® p-value format of "< 0.0001" or "> 0.9999" will be reported.
- Unless otherwise noted, the denominator for percentages is the number of subjects in the applicable analysis population and treatment group.
- If the frequency for a particular table cell is zero, then "0", properly aligned, will be displayed (i.e. "0 (0.0%)" will not be displayed.)
- Non-numeric values: Where variables are recorded using < (e.g., "< 10" or "≤ 10") the numeric portion of the result will be used (e.g., < 10 and ≤ 10 becomes 10) for summary; where variables are recorded using > (e.g., "> 10" or " ≥ 10") the numeric portion of the result will be used (e.g. > 10 and ≥ 10 become 10) for summary; the actual recorded results, (e.g. "< 10" or "> 10") will appear in listings.

#### 14.1. GENERAL CONSIDERATIONS

A separate SAS program will be created for each output.

1007779

- Output files will be delivered in Word format.
- Numbering of TFLs will follow ICH E3 guidance

## 14.2. TABLE, LISTING, AND FIGURE FORMAT

#### 14.2.1. General

- All TLFs will be produced in landscape format, unless otherwise specified.
- All TLFs will be produced using the Courier New font, size 9
- The data displays for all TLFs will have a minimum 1-inch margin on all 4 sides.
- Headers and footers for figures will be in Courier New font, size 9.
- Legends will be used for all figures with more than 1 variable, group, or item displayed.
- TLFs will be in black and white (no color), unless otherwise specified
- Specialized text styles, such as bolding, italics, borders, shading, and superscripted and subscripted text, will not be used in the TLFs, unless otherwise specified. On some occasions, superscripts 1, 2, or 3 may be used (see below).
- Only standard keyboard characters will be used in the TLFs. Special characters, such as non-printable control characters, printer-specific, or font-specific characters, will not be used. Hexadecimal-derived characters will be used, where possible, if they are appropriate to help display math symbols (e.g., µ). Certain subscripts and superscripts (e.g., cm2, Cmax) will be employed on a case-by-case basis.
- Mixed case will be used for all titles, footnotes, column headers, and programmer-supplied formats, as appropriate.

#### 14.2.2. Headers

- All output should have the following header at the top left of each page:
  - Theracos Sub. LLC
  - Protocol Number: THR-1442-C-423
- Draft or Final in top right corner.
- All output should have Page n of N at the top of each page. TLFs should be internally paginated in relation to the total length (i.e., the page number should appear sequentially as page n of N, where N is the total number of pages in the table).
- The date output was generated should appear along with the program name as a footer on each page.

1007779

## 14.2.3. Display Titles

• Each TLF should be identified by the designation and a numeral. (i.e., Table 14.1.1). ICH E3 numbering is strongly recommended but sponsor preferences should be obtained prior to final determination. A decimal system (x.y and x.y.z) should be used to identify TLFs with related contents. The title is centered. The analysis set should be identified on the line immediately following the title. The title and table designation are single spaced. A solid line spanning the margins will separate the display titles from the column headers. There will be 1 blank line between the last title and the solid line.

Table x.y.z
First Line of Title
Second Line of Title if Needed
ITT Analysis Set

#### 14.2.4. Column Headers

- Column headings should be displayed immediately below the solid line described above in initial upper-case characters.
- In the case of efficacy tables, the variable (or characteristic) column will be on the far left followed by the treatment group columns and total column (if applicable). P-values will be presented in a separate comparison column (if applicable).
- For numeric variables, include "unit" in column or row heading when appropriate.
- Analysis set sizes will be presented for each treatment group in the column heading as (N=xx) (or in the row headings if applicable). This is distinct from the 'n' used for the descriptive statistics representing the number of subjects in the analysis set.
- The order of treatments in the tables and listings will be active treatment first, then active control, followed by a total column (if applicable).

#### 14.2.5. Body of the Data Display

#### 14.2.5.1. General Conventions

Data in columns of a table or listing should be formatted as follows:

- alphanumeric values are left-justified;
- whole numbers (e.g., counts) are right-justified; and
- numbers containing fractional portions are decimal aligned.

1007779

#### 14.2.5.2. Table Conventions

- Units will be included where available
- If the categories of a parameter are ordered, then all categories between the maximum and minimum category should be presented in the table, even if n=0 for all treatment groups in a given category that is between the minimum and maximum level for that parameter. For example, the frequency distribution for symptom severity would appear as:

| Severity | N |
|----------|---|
| Rating | |
| severe | 0 |
| moderate | 8 |
| mild | 3 |

Where percentages are presented in these tables, zero percentages will not be presented and so any counts of 0 will be presented as 0 and not as 0 (0%).

- If the categories are not ordered (e.g., Medical History, Reasons for Discontinuation from the Study, etc.), then only those categories for which there is at least 1 subject represented in 1 or more groups should be included.
- An Unknown or Missing category should be added to any parameter for which information is not available for 1 or more subjects.
- Unless otherwise specified, the estimated mean and median for a set of values should be printed out to 1 more significant digit than the original values, and standard deviations should be printed out to 2 more significant digits than the original values. The minimum and maximum should report the same significant digits as the original values. For example, for systolic blood pressure:

| n | XX |
|---------|-------|
| Mean | XXX.X |
| SD | X.XX |
| Q1 | XXX.X |
| Median | XXX.X |
| Q3 | XXX.X |
| Minimum | XXX |
| Maximum | XXX |

- P-values should be output in the format: "0.xxxx", where xxxx is the value rounded to 4 decimal places. Any p-value less than 0.0001 will be presented as <0.0001. If the p-value is returned as >0.9999 then present as >0.9999
- Percentage values should be printed to one decimal place, in parentheses with no spaces, one space after the count (e.g., 7 (12.8%), 13 (5.4%)). If the rounded percentage is 0.0, display as '<0.1'. Unless otherwise noted, for all percentages, the number of subjects in the analysis set for the treatment group who have an observation will be the denominator. Percentages after zero counts should not be

1007779

- displayed and percentages equating to 100% should be presented as 100%, without any decimal places.
- Tabular display of data for concomitant and rescue medications should be presented by treatment class with the highest occurrence in the total column in decreasing order. Tabular display of data for medical history and adverse event data should be presented by the SOC using descending order. Within the drug class and SOC, medical history (by preferred term), drugs (by ATC2 code), and adverse events (by preferred term) should be displayed in decreasing order in the total column. If incidence for more than 1 term is identical, they should then be sorted alphabetically. Missing descriptive statistics which cannot be estimated should be reported as "-".
- The percentage of subjects is normally calculated as a proportion of the number of subjects assessed in the relevant treatment group (or overall) for the analysis set presented. However, careful consideration is required in many instances due to the complicated nature of selecting the denominator, usually the appropriate number of subjects exposed. Describe details of this in footnotes or programming notes.
- For categorical summaries (number and percentage of subjects) where a subject can be included in more than one category, describe in a footnote or programming note if the subject should be included in the summary statistics for all relevant categories or just 1 category and the criteria for selecting the criteria.
- Where a category with a subheading (such as system organ class) has to be split over more than one page, output the subheading followed by "(cont)" at the top of each subsequent page. The overall summary statistics for the subheading should only be output on the first relevant page.

#### 14.2.5.3. Listing Conventions

- Listings will be sorted for presentation in order of treatment groups as above, subject number, visit/collection day, and visit/collection time.
- Missing data should be represented on subject listings as either a hyphen ("-") with a corresponding footnote ("- = unknown or not evaluated"), or as "N/A", with the footnote "N/A = not applicable", whichever is appropriate.
- Dates should be printed in SAS® DATE9.format ("ddMMMyyyy": 01JUL2000). Missing portions of dates should be represented on subject listings as dashes (--JUL2000).
   Dates that are missing because they are not applicable for the subject are output as "N/A", unless otherwise specified.
- All observed time values must be presented using a 24-hour clock HH:MM or HH:MM:SS format (e.g., 11:26:45, or 11:26). Time will only be reported if it was measured as part of the study.
- Units will be included where available

1007779

#### 14.2.5.4. Figure Conventions

 Unless otherwise specified, for all figures, study visits will be displayed on the X-axis and endpoint (e.g., treatment mean change from Baseline) values will be displayed on the Y-axis.

#### 14.2.6. Footnotes

- A solid line spanning the margins will separate the body of the data display from the footnotes.
- All footnotes will be left justified with single-line spacing immediately below the solid line underneath the data display.
- Footnotes should always begin with "Note:" if an informational footnote, or 1, 2, 3, etc. if a reference footnote. Each new footnote should start on a new line where possible.
- Subject specific footnotes should be avoided, where possible.
- Footnotes will be used sparingly and must add value to the table, figure, or data listing. If more than six lines of footnotes are planned, then a cover page may be used to display footnotes, and only those essential to comprehension of the data will be repeated on each page.
- The last line of the footnote section will be a standard source line that indicates the name of the program used to produce the data display, date the program was run, and the listing source (i.e., 'Program: myprogram.sas Listing source: 16.x.y.z').

# 15. QUALITY CONTROL

SAS programs are developed to produce clinical trial output such as analysis data sets, summary tables, data listings, figures or statistical analyses. INC Research SOP 03.010 and 03.013 provide an overview of the development of such SAS programs.

INC Research SOP 03.009 describes the quality control procedures that are performed for all SAS programs and output. Quality control is defined here as the operational techniques and activities undertaken to verify that the SAS programs produce the proper clinical trial output by checking for their logic, efficiency and commenting and by review of the produced output.

1007779

- 16. INDEX OF TABLES
- 17. INDEX OF FIGURES
- 18. INDEX OF LISTINGS
- 19. MOCK-UPS

Attachment 1: Planned Table Shells

Attachment 2: Planned Listing Shells

Attachment 3: Planned Figure Shells

# 20. APPENDICES